CLINICAL TRIAL: NCT03385902
Title: Impact on Mortality of Timing of Dialysis Initiation in Patients With End-stage Renal Disease by a Novel Assessment Based on Fuzzy Mathematics
Brief Title: Assessment of Dialysis Initiation by a Fuzzy Mathematics Equation
Acronym: ADIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Chinese PLA General Hospital (Other); Fudan University (Other); RenJi Hospital (Other); Guangdong Provincial People's Hospital (Other); Beijing Friendship Hospital (Other); Huashan Hospital (Other); West China Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); General hospital of benxi iron and steel co. (Unknown); Dalian Municipal Central Hospital (Other); An Steel Group Hospital (Unknown); The First Affiliated Hospital of the Fourth Military Medical University (Other); General Hospital of Mining Industry Group Fuxin (Unknown); Affiliated Zhongshan Hospital of Dalian University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); General Hospital of Ningxia Medical University (Other); LanZhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Henan Provincial People's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Hospital of China Medical University (Other); Central Hospital Affiliated to Shenyang Medical Collage (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YJ-KY-2017-119
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease
Keywords: end-stage renal disease; timing of dialysis initiation; hemodialysis; fuzzy mathematics; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimal start dialysis group (Experimental): The DIFE will be used as the assessment of initiation time of dialysis. Patients in this group will start dialysis when their results of the DIFE reaching to 30-35, which defined as the optimal start time.
  Interventions: Other: optimal start time
- late start dialysis group (Active Comparator): the DIFE will be used as the assessment of initiation time of dialysis. Patients in this group will start dialysis when their results of the DIFE less than 30, which defined as late start time.
  Interventions: Other: late start time

INTERVENTIONS:
Other: optimal start time — patients will start hemodialysis when their DIFE reach 35, and can not wait if the DIFE decline to 30.
  Arms: optimal start dialysis group
Other: late start time — patients will start hemodialysis when their DIFE less than 30
  Arms: late start dialysis group

SUMMARY:
The purpose of this study is to evaluate the impact of the optimal and late initiation of dialysis on the mortality and quality of life in end-stage renal disease (ESRD) patients by the Dialysis Initiation based on Fuzzy mathematics Equation (DIFE), which is a novel equation for the assessment of timing of dialysis initiation established by Fuzzy mathematics.

DETAILED DESCRIPTION:
The optimal time of dialysis initiation is still controversial. Estimated glomerular filtration rate (eGFR) which is now widely used as the assessment of timing of dialysis is lack of specificity. Some clinical factors such as heart failure, volume overload, malnutrition also determine the dialysis time. But these subjective judgements do not have a standard. So there is no quantitative assessment of timing of dialysis initiation. The research team developed a novel equation named DIFE (Dialysis Initiation based on Fuzzy mathematics Equation) with data from a retrospective multicenter cohort by fuzzy mathematical methods to combine these clinical factors and lab indexes. The DIFE was confirmed to be more accurate and convenient to use in clinical practice than eGFR only at the assessment of dialysis initiation time in the internal validation. For further validation of the DIFE, the team will conduct a multicenter randomized controlled trial. Patients who need hemodialysis will be randomized to optimal start dailysis group or late start dailysis group by the assessment of the DIFE. Based on the comparison of the two groups, this trial will provide evidence for the optimal timing of dialysis initiation in patients with end-stage renal disease by the DIFE.

ELIGIBILITY:
Inclusion Criteria:

* Have progressive chronic kidney disease with an eGFR less than 15 ml/min/1.73m2 and a DIFE between 30-35
* Expected to commence maintenance hemodialysis as their renal replacement treatment
* Agreeable to randomization

Exclusion Criteria:

* Acute kidney injury (AKI) or AKI on chronic kidney disease (CKD)
* With the primary disease of systemic lupus erythematosus (SLE) or systemic vasculitis
* Have received or planning to receive a kidney transplant or peritoneal dialysis during the study
* Has a recently diagnosed cancer that was likely to affect survival (except for the following cases: the cancer has been confirmed to be cured or relieved for over 5 years, have had the radical resection for the basal cell carcinoma or squamous carcinoma of skin or carcinoma in-situ of any part of the body )
* Hepatocirrhosis
* Positive test of Human Immunodeficiency Virus (HIV), the hepatitis B virus antigen (HBsAg) or anti-hepatitis C virus antibody (HCV Ab)
* Acute infection within 1 month
* Bad habit which is difficult to withdrawal such as alcohol abuse
* Poor compliance and could not be treated according to the protocol
* Being pregnant, nursing or having a plan for pregnancy
* Life expectancy less than 1 year
* The investigator confirm that should not enroll in the study with any other cases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2018-04-14 (Actual); Primary Completion 2023-08-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | from the date of enrollment until the end of study, assessed up to 3 years
  proportion of patients who die from any cause
cerebro-cardiovascular mortality | 3 years, from the date of enrollment until the end of study
  proportion of patients who die from cerebro-cardiovascular disease

SECONDARY OUTCOMES:
cerebro-cardiovascular events | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  proportion of patients who suffer from cardiovascular events, which include nonfatal myocardial infarction, nonfatal stroke, transient ischemic attack,new-onset angina, acute heart failure or severe arrhythmia.
hospitalization | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  proportion of patients admitted to hospital
Nutrition assessment | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  assess the patient's nutritional status by subjective global assessment (SGA) assessment and serum albumin level
the change of quality of life | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  use short form-36 reported by the patients to assess the patient's quality of life
Medical cost | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  the cost by the patient, family and insurance during treatment
Hemodialysis complications | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  the proportion of patients who suffer from hemodialysis complications including blood assess revise, assess infection, severe fluid and electrolyte disorders
cognitive dysfunction | from the date of enrollment until the date of death from any cause, or the end of study, which ever came first, assessed up to 3 years
  assess cognitive dysfunction by Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Lin, MD， PhD, Study Director — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- the First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper BA, Branley P, Bulfone L, Collins JF, Craig JC, Fraenkel MB, Harris A, Johnson DW, Kesselhut J, Li JJ, Luxton G, Pilmore A, Tiller DJ, Harris DC, Pollock CA; IDEAL Study. A randomized, controlled trial of early versus late initiation of dialysis. N Engl J Med. 2010 Aug 12;363(7):609-19. doi: 10.1056/NEJMoa1000552. Epub 2010 Jun 27. PMID 20581422
- [Result] Crews DC, Scialla JJ, Boulware LE, Navaneethan SD, Nally JV Jr, Liu X, Arrigain S, Schold JD, Ephraim PL, Jolly SE, Sozio SM, Michels WM, Miskulin DC, Tangri N, Shafi T, Wu AW, Bandeen-Roche K; DEcIDE Network Patient Outcomes in End Stage Renal Disease Study Investigators. Comparative effectiveness of early versus conventional timing of dialysis initiation in advanced CKD. Am J Kidney Dis. 2014 May;63(5):806-15. doi: 10.1053/j.ajkd.2013.12.010. Epub 2014 Feb 6. PMID 24508475
- [Result] Susantitaphong P, Altamimi S, Ashkar M, Balk EM, Stel VS, Wright S, Jaber BL. GFR at initiation of dialysis and mortality in CKD: a meta-analysis. Am J Kidney Dis. 2012 Jun;59(6):829-40. doi: 10.1053/j.ajkd.2012.01.015. Epub 2012 Apr 1. PMID 22465328
- [Result] Nesrallah GE, Mustafa RA, Clark WF, Bass A, Barnieh L, Hemmelgarn BR, Klarenbach S, Quinn RR, Hiremath S, Ravani P, Sood MM, Moist LM; Canadian Society of Nephrology. Canadian Society of Nephrology 2014 clinical practice guideline for timing the initiation of chronic dialysis. CMAJ. 2014 Feb 4;186(2):112-7. doi: 10.1503/cmaj.130363. No abstract available. PMID 24492525
- [Result] Sood MM, Komenda P, Rigatto C, Hiebert B, Tangri N. The association of eGFR reporting with the timing of dialysis initiation. J Am Soc Nephrol. 2014 Sep;25(9):2097-104. doi: 10.1681/ASN.2013090953. Epub 2014 Mar 20. PMID 24652801
- [Result] Hwang SJ, Yang WC, Lin MY, Mau LW, Chen HC; Taiwan Society of Nephrology. Impact of the clinical conditions at dialysis initiation on mortality in incident haemodialysis patients: a national cohort study in Taiwan. Nephrol Dial Transplant. 2010 Aug;25(8):2616-24. doi: 10.1093/ndt/gfq308. Epub 2010 Jun 2. PMID 20519231
- [Derived] Chen J, Liu Y, Chen X, Sun X, Li W, Yang W, Li P, Sun X, Wang D, Jiang H, Shi W, Liu W, Fu P, Ding X, Chang M, Liu S, Yang X, Cao N, Chen M, Ni Z, Chen J, Sun S, Liang X, Wang H, He Y, Gao B, Wang J, Hao L, Liu J, Li S, He Q, Liu H, Yi N, Shao F, Jiao J, Ma Y, Yao L, Sun Y, Li D, Szczech L, Fang M, Odeh Z, Lin H. Assessment of dialysis initiation by a fuzzy mathematics equation (ADIFE): a study protocol for a randomised controlled trial. BMJ Open. 2019 Sep 8;9(9):e023162. doi: 10.1136/bmjopen-2018-023162. PMID 31501092